CLINICAL TRIAL: NCT03080831
Title: TOnicity of Perioperative Maintenance SoluTions - Part 1: Thoracic Surgery
Brief Title: TOnicity of Perioperative Maintenance SoluTions
Acronym: TOPMAST-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Niels Van Regenmortel (Other)
Responsible Party: Sponsor-Investigator, Niels Van Regenmortel, Dr., University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 17/4/34
Record Dates: First submitted 2017-02-19; First posted 2017-03-15 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Thoracic Diseases; Water-Electrolyte Imbalance; Fluid Overload; Fluid Retention; Sodium Disorder; Potassium Disorders; Chloride Disorder
Keywords: Maintenance Fluid Therapy
MeSH Terms: conditions — Thoracic Diseases; Water-Electrolyte Imbalance; Edema | interventions — Glucose; Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study fluids blinded using opaque bags
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NaCl 0.9% in Glucose 5% + 40mmol/L Potassium (Active Comparator)
  Interventions: Drug: NaCl 0.9% in Glucose 5% + 40mmol/L Potassium
- Glucion 5% (Active Comparator)
  Interventions: Drug: Glucion 5%

INTERVENTIONS:
Drug: NaCl 0.9% in Glucose 5% + 40mmol/L Potassium — Study fluid used at maintenance rate of 27 mmol per kg of body weight per day from beginning of surgery until end of study.
  Arms: NaCl 0.9% in Glucose 5% + 40mmol/L Potassium
Drug: Glucion 5% — Study fluid used at maintenance rate of 27 mmol per kg of body weight per day from beginning of surgery until end of study.
  Arms: Glucion 5%

SUMMARY:
Prospective randomized double blind phase IV trial studying the efficacy and safety of the tonicity of two different perioperative maintenance solutions: an isotonic solution containing NaCl 0.9 in glucose 5% with an added 40 mmol/L of potassium or a commercially available premixed solution (Glucion 5%) containing a.o. 54 mmol/L of sodium and 26 mmol/L of potassium. Both solutions are administered at 27 mL/kg of ideal body weight, as recommended by current guidelines (NICE 174) and both solutions are widely used in daily clinical practice. The primary hypothesis is that isotonic maintenance solutions lead to more fluid retention than hypotonic fluids. Metabolism of both solutions is assessed by sequential analysis of urine and serum and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 y.o.)
* Undergoing elective lung resection (wedge resection, segmental resection, (bi)lobectomy, but not pneumonectomy) via thoracotomy or video- or robot assisted (VATS, RATS)
* Normal renal function (eGFR >60 ml/min/1.73m² (CKD-EPI))

Exclusion Criteria:

* Under chronic treatment with diuretics or desmopressin
* Heart failure (NYHA III-IV)
* Liver Failure
* Brittle diabetes mellitus
* Neurological contra-indication for hypotonic fluids
* SIADH or hyponatremia <130 or > 150 mmol/L at preoperative assessment
* Hyperkalemia > 5 mmol/L at preoperative assessment
* Under treatment with artificial nutrition (enteral or parenteral)
* Pregnancy

Additional pre-defined exclusion after initial inclusion

* Massive perioperative transfusion or intraoperative resuscitation of +2.5L of crystalloids/colloids
* Absence of admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Fluid balance | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery)
  Difference between all fluid intake and output

SECONDARY OUTCOMES:
Resuscitation Fluids | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery)
  The cumulative amount of additional (resuscitation) fluids during the study period
Vasopressor Use | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery)
  The cumulative amount of vasopressors during the study period
Physiological Mechanisms: Aldosterone level | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Change from baseline aldosterone level at start of surgery
Physiological Mechanisms: Fractional Excretion of Sodium | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Change from baseline FeNa at start of surgery
Electrolyte Homeostasis and Disorders: Sodium | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean sodium level and change from baseline. Occurrence of hypo and hypernatremia.
Electrolyte Homeostasis and Disorders: Potassium | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean potassium level and change from baseline. Occurrence of hypo and hyperpotassemia.
Electrolyte Homeostasis and Disorders: Chloride | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean chloride level and change from baseline. Occurrence of hypo and hyperchloremia.
Electrolyte Homeostasis and Disorders: Strong Ion Difference | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean SID level and change from baseline.
Electrolyte Homeostasis and Disorders: Phosphate | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean phosphate level and change from baseline. Occurrence of hypo and hyperphosphatemia.
Electrolyte Homeostasis and Disorders: Calcium | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean calcium level and change from baseline. Occurrence of hypo and hypercalcemia.
Clinical Endpoints: paO2/FiO2 | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery) - Assessments at fixed time points.
  Mean postoperative paO2/FiO2
Clinical Endpoints: occurrence of de novo atrial fibrillation | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery). Continuous assessment.
  occurrence of de novo atrial fibrillation (Y/N)
Clinical Endpoints: occurrence of acute kidney injury (AKI) | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery). Continuous assessment.
  AKI according to RIFLE-score creatinine and urine R-I-F)
Sodium balance | From start of surgery until end of study, defined as one of the following (1) discharge from ICU (2) 8AM on third postoperative day (maximum: up to 72h after start of surgery).
  Sodium balance (total in vs out) at end of study, assessed by urine collection.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Antwerp, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data available on reasonable request

REFERENCES:
- [Background] Lobo DN, Bostock KA, Neal KR, Perkins AC, Rowlands BJ, Allison SP. Effect of salt and water balance on recovery of gastrointestinal function after elective colonic resection: a randomised controlled trial. Lancet. 2002 May 25;359(9320):1812-8. doi: 10.1016/S0140-6736(02)08711-1. PMID 12044376
- [Background] Moritz ML, Ayus JC. Maintenance Intravenous Fluids in Acutely Ill Patients. N Engl J Med. 2015 Oct;373(14):1350-60. doi: 10.1056/NEJMra1412877. No abstract available. PMID 26422725
- See also: NICE guideline on Intravenous Fluid Therapy in Adults in Hospital — http://guidance.nice.org.uk/CG174
- See also: GIFTASUP guidelines — http://www.bapen.org.uk/pdfs/bapen_pubs/giftasup.pdf